CLINICAL TRIAL: NCT05546840
Title: Reporting Usual Physiotherapy Care in Stroke Survivors in Catalonia
Acronym: UsualPTCare
Status: Completed | Type: Observational
Sponsor: Universitat de Lleida (Other)
Collaborators: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Maria Masbernat-Almenara, Principal Investigator, Universitat de Lleida
Other Study IDs: P22/000
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: stroke; Physiotherapy; rehabilitation; catalonia; usual care
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke is one of the major leading causes of death and disability globally and presents a high interest of research around all its branches, including rehabilitation. There are published recommendations and clinical guidelines to guide the care of stroke patients with regard to physical therapy. However, the status of current clinical practice is unknown.

This study aims to identify and describe the therapeutic approaches most used by physiotherapists in Catalonia in the care of stroke survivors in different phases of evolution.

An observational study will be carried out through an anonymous survey of physiotherapists in Catalonia. Through the College of Physiotherapists of Catalonia, all members will be invited to answer a survey on current clinical practice in the care of stroke survivors. The survey will collect data related to the physiotherapist's training and experience, the most frequently used therapeutic approaches, user profiles and institutions. It is intended to collect the data between October 2022 and February 2023. The data will be analyzed by the team of researchers

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapists who are currently working in Catalonia with patients who have suffered a stroke.

Exclusion Criteria:

* Physiotherapists do not currently work with at least one stroke patient

Ages: 22 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Physiotherapists specialized in neurorehabilitation who in their day to day care for patients with stroke.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Demographic data | Day 1
  Gender, Age, postal code, completion of degree studies, formation in neurology
Specific formation in neurology | Day 1
  CV information
Neurorehabilitation experience | Day 1
  Years of experience, work place,
Multidisciplinary team | Day 1
  Multidisciplinary co-workers such as Physical therapists, occupational therapists, medical doctors, psychologists
Therapeutic intervention | Day 1
  Sessions, doses, type of patients, type of intervention, approaches,
Individual therapy | Day 1
  Doses, time,
Group Therapy | Day 1
  Doses, Time
Therapy | Day 1
  Doses, time

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lleida, Lleida, Spain

REFERENCES:
- [Derived] Masbernat-Almenara M, Hervas SP, Fernandez-Lago H, Gonzalez-Hoelling S, Salgueiro C, Cabanas-Valdes R. Mapping Physiotherapy Approaches for Stroke Survivors in Catalonia: A Cross-Sectional Study. Rev Neurol. 2025 Jun 16;80(5):37316. doi: 10.31083/RN37316. PMID 40613408